CLINICAL TRIAL: NCT01766453
Title: Utility of a Culturally Relevant or a Standard Exercise Program to Reduce Visceral Adipose Tissue and Cardiovascular Disease Risk in Abdominally Obese Postmenopausal South Asian Women
Brief Title: South Asian Yoga and Exercise Trial
Acronym: SAYET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Scott Lear, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SFU
Record Dates: First submitted 2012-12-11; First posted 2013-01-11 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: South Asian; Cardiovascular; Exercise; Obesity; Visceral Adipose Tissue
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non exercise control (No Intervention): Non exercise control will undergo baseline testing and follow up testing but will not participate in an exercise intervention.
- Standard Exercise (Experimental): The standard exercise group will attend exercise sessions under the supervision of a Certified Personal Trainer. Intensity will increase every four weeks by 10% from 50-80% of maximal heart rate to ensure that exercise is progressive in nature. Participants will be provided with a heart rate monitor during their exercise sessions and have the option to perform the aerobic training on a treadmill, upright bike, elliptical machine or recumbent bike as long as heart rate is kept within the prescribed training intensity. Intensity, duration, resting and exercise heart rates will be recorded for each exercise session for the duration of the intervention to ensure compliance to the exercise program.
  Interventions: Behavioral: Standard Exercise
- Bhangra Dance Exercise (Experimental): Bhangra dance classes taught be a certified instructor progressing in difficulty over the 12 week period. Bhangra dance is an Indian folk dance that consists of jumping and kicking of a high intensity. This group will attend exercise sessions under the supervision of a Bhangra Dance Instructor. The intensity of bhangra dance will be tracked through heart rate monitors worn by participants.
  Interventions: Behavioral: Bhangra dance exercise

INTERVENTIONS:
Behavioral: Standard Exercise — Aerobic exercise with a progressive increase in intensity over 12 weeks.
  Arms: Standard Exercise
Behavioral: Bhangra dance exercise — Bhangra Dance classes taught by an instructor.
  Arms: Bhangra Dance Exercise

SUMMARY:
South Asians have one of the highest rates of heart disease of all populations and a unique and deleterious obesity phenotype of increased body fat and inner-abdominal compared to those of European background. We have subsequently identified that this unique phenotype accounts for much of the increased heart disease risk in South Asians, with the greater amounts of inner abdominal fat being particularly implicated. In addition, South Asians in Canada have substantially lower levels of leisure-time physical activity.

At present, we do not know the answers to the following questions:

1. Is a conventional (standard) physical activity program that has proven effective at reducing inner abdominal fat and heart disease risk factors in populations of European background be effective in South Asians?
2. Is an alternative physical activity program commonly practiced by South Asians (such as bhangra dance) be effective at reducing inner abdominal fat and heart disease risk factors in South Asians? In this study, we will perform a randomized controlled trial of three conditions-gym-based standard exercise program (SE),bhangra dance exercise program (BE) and non-exercise control (NE).We will recruit 75 post-menopausal South Asian women with abdominal obesity and assign them randomly to one of the three groups (25 per group).

We anticipate that both the SE and BE programs will be superior to the NE group in terms of reducing VAT and CVD risk factors. Such findings will demonstrate that exercise is an effective method that favourably modifies the obesity phenotype of excess VAT in South Asians, and should be central to health promotion and disease prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal South Asian women defined as not menstruating for the previous 12 consecutive months as assessed by self report
* Waist circumference >80 cm (women), as identified as South Asian cut offs by International Diabetes Federation109
* Able to read and write and understand English
* Previously sedentary (<150 minutes of physical activity per week as assessed by accelerometry)
* Weight stable (<2kg of weight change over the past 6 weeks)

Exclusion Criteria:

* Taking medication that may affect study outcomes (lipid-lowering, antihypertensive, or hypoglycemic medications)
* Unable to provide informed consent
* Individuals > 136 kg (physical limitation of DXA scanner table)
* Smokers (given the confounding association between smoking and adiposity)
* Unable to participate in exercise sessions due to physical limitations or contra-indications to regular exercise as indicated on the baseline maximal exercise stress test
* Individuals with known CVD or other known comorbidities (HIV, immune compromised condition, type 1 or 2 diabetes mellitus)
* Another member of the household already participating in study

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visceral adipose tissue | 12 weeks
  Visceral adipose tissue will be assessed with multi-slice computed tomography

SECONDARY OUTCOMES:
Cardiometabolic risk factors | 12 weeks
  Blood will be drawn and assessed for lipids, glucose, insulin, CRP, adiponectin and ALT
Body Composition | 12 weeks
  DEXA scans will be used to assess body fat distribution and lean body mass
Maximal Aerobic Fitness | 12 weeks
  A Bruce protocol treadmill test with metabolic data will be used to assess aerobic fitness

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Lear, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- Simon Fraser University, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Lesser IA, Singer J, Hoogbruin A, Mackey DC, Katzmarzyk PT, Sohal P, Leipsic J, Lear SA. Effectiveness of Exercise on Visceral Adipose Tissue in Older South Asian Women. Med Sci Sports Exerc. 2016 Jul;48(7):1371-8. doi: 10.1249/MSS.0000000000000906. PMID 26909531